CLINICAL TRIAL: NCT00160966
Title: Prospective Randomized Study to Characterize Risk Factors of Polyomavirus-related Transplant Nephropathy and the Impact of Three Immunosuppressive Regimens on Nephropathy Incidence
Brief Title: Impact of Immunosuppressive Regimens on Polyomavirus-related Transplant Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Heidelberg University (Other); Hoffmann-La Roche (Industry); Astellas Pharma Inc (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Rolf Weimer, Prof. Dr., University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTx-PV-002
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-01

CONDITIONS: Polyomavirus Infections
Keywords: kidney transplantation; polyoma virus associated transplant nephropathy; tacrolimus; mycophenolate mofetil; everolimus; cyclosporin A; BK virus PCR; viruria screening; BK polyomavirus; immunosuppression
MeSH Terms: conditions — Polyomavirus Infections | interventions — Cyclosporine; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Immunosuppression with Ciclosporin and Mycophenolate-mofetil; Ciclosporin treatment being started at the latest at day 4 after transplantation with 7 mg/kg body weight daily administered every 8 hours until the target trough level of 300 µg/l was reached. Then it was administered twice daily with daily monitoring of trough levels. The target trough level was lowered to 200 µg/l 1 month after transplantation. Thereafter dosage and target trough levels were adjusted at the investigators discretion. Mycophenolate-mofetil was started previous to transplantation procedure with a starting dosage of 3 g/day administered twice daily. Once ciclosporin was entered into the therapy-scheme Mycophenolate-mofetil dosage was reduced to 2 g/daily. The therapy was controlled by measuring of trough levels with a target trough level exceeding 1 µg/ml. The dosage was adjusted at the investigators discretion.
  Interventions: Drug: Ciclosporin and Mycophenolate-mofetil
- 2 (Active Comparator): Immunosuppression with Tacrolimus and Mycophenolate-mofetil Mycophenolate-mofetil was started previous to transplantation procedure with a starting dosage of 3 g/day administered twice daily. Once tacrolimus was entered into the therapy-scheme Mycophenolate-mofetil dosage was reduced to 2 g/daily. The therapy was controlled by measuring of trough levels with a target trough level exceeding 1 µg/ml. The dosage was adjusted to clinical signs of overimmunosuppression (infections) or intolerance (mainly gastrointestinal side effects) or rejections.
  Interventions: Drug: Tacrolimus and Mycophenolate-mofetil
- 3 (Active Comparator): Immunosuppression with Tacrolimus and Mycophenolate-mofetil with change from Mycophenolate-mofetil to Everolimus after completion of posttransplant wound healing
  Interventions: Drug: Tacrolimus and Mycophenolate-mofetil with change from Mycophenolate-mofetil to Everolimus

INTERVENTIONS:
Drug: Ciclosporin and Mycophenolate-mofetil — according to the Giessen protocol
  Arms: 1
Drug: Tacrolimus and Mycophenolate-mofetil — according to Giessen protocol
  Arms: 2
Drug: Tacrolimus and Mycophenolate-mofetil with change from Mycophenolate-mofetil to Everolimus — according to Giessen protocol
  Arms: 3

SUMMARY:
The aim of this study is to characterize and evaluate risk factors of polyomavirus nephropathy (PVN) including the impact of three immunosuppressive regimens.

DETAILED DESCRIPTION:
Polyomavirus nephropathy (PVN) is an emerging cause of renal transplant loss. Until now the risk factors of PVN are poorly understood. Tacrolimus (Tacr) and mycophenolate mofetil (MMF) are thought to be associated with a higher risk of developing PVN. However, the way in which Tacr or MMF might enhance the susceptibility for PVN remains largely unknown. In this prospective study we will analyze whether differences in immune-reactivity patterns (Th1, Th2, B cell and monocyte responses, sCD30, immunoregulatory antibodies) of renal transplant patients induced by different immunosuppressive regimens (cyclosporine A [CsA]/MMF, Tacr/MMF, Tacr/MMF with conversion to Tacr/Everolimus [ERL]) or by cytokine promoter gene polymorphisms may account for the different risks of developing PVN.

Comparison(s): renal transplant recipients stratified according to their relative immunological risk (group 1: low risk (primary recipients without pre-immunization [PRA < 5%]); group 2: moderate risk (group 2a: primary recipients with low pre-immunization [PRA 6-20%]; group 2b: re-transplanted patients); group 3: very high risk (re-transplanted patients with a history of vascular rejection or recipients of a first graft with high pre-immunization [PRA > 20%]) randomized to be treated with one of three immunosuppressive regimens (CsA/MMF, Tacr/MMF, Tacr/MMF with subsequent conversion to Tacr/ERL).

ELIGIBILITY:
Inclusion Criteria:

* Cadaver kidney and living donor kidney transplant recipients
* Primary, secondary, and tertiary transplant recipients
* Pre-immunized and not pre-immunized transplant recipients
* Age > 18 years

Exclusion Criteria:

* Contraindications against administration of one of the four study drugs
* History of severe gastrointestinal morbidity
* Age < 18 years
* Pregnant or breast feeding women
* Rejection of effective contraceptive methods with young women
* Combined kidney and islet cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
incidence of polyomavirus associated transplant nephropathy (PVN) | 2 years posttransplant
incidence of polyoma viremia | 2 years posttransplant
urine polyomavirus concentration within the first two years post-transplant | 2 years posttransplant

SECONDARY OUTCOMES:
patients' and grafts' survival | 2 years posttransplant
incidence of acute rejections | 2 years posttransplant
transplant function 1 and 2 years post-transplant | 2 years posttransplant
comparison of urine cytology and polymerase chain reaction (PCR) quantitative data regarding diagnosis of PVN | 2 years posttransplant
predictive value of immune parameters prognostically relevant for acute or chronic rejection | 2 years posttransplant
side effects of immunosuppressive drugs | 2 years posttransplant

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Weimer, Prof., MD, Principal Investigator — University Giessen, Internal Medicine
Locations (1):
- Department of Internal Medicine, University of Giessen, Giessen, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of all participants will be made available within 1 year of study completion.

REFERENCES:
- [Background] Andrews CA, Shah KV, Daniel RW, Hirsch MS, Rubin RH. A serological investigation of BK virus and JC virus infections in recipients of renal allografts. J Infect Dis. 1988 Jul;158(1):176-81. doi: 10.1093/infdis/158.1.176. PMID 2839580
- [Background] Barri YM, Ahmad I, Ketel BL, Barone GW, Walker PD, Bonsib SM, Abul-Ezz SR. Polyoma viral infection in renal transplantation: the role of immunosuppressive therapy. Clin Transplant. 2001 Aug;15(4):240-6. doi: 10.1034/j.1399-0012.2001.150404.x. PMID 11683817
- [Background] Nickeleit V, Hirsch HH, Zeiler M, Gudat F, Prince O, Thiel G, Mihatsch MJ. BK-virus nephropathy in renal transplants-tubular necrosis, MHC-class II expression and rejection in a puzzling game. Nephrol Dial Transplant. 2000 Mar;15(3):324-32. doi: 10.1093/ndt/15.3.324. PMID 10692517
- [Background] Hirsch HH, Knowles W, Dickenmann M, Passweg J, Klimkait T, Mihatsch MJ, Steiger J. Prospective study of polyomavirus type BK replication and nephropathy in renal-transplant recipients. N Engl J Med. 2002 Aug 15;347(7):488-96. doi: 10.1056/NEJMoa020439. PMID 12181403
- [Background] Hirsch HH. Polyomavirus BK nephropathy: a (re-)emerging complication in renal transplantation. Am J Transplant. 2002 Jan;2(1):25-30. doi: 10.1034/j.1600-6143.2002.020106.x. PMID 12095052
- [Background] Hirsch HH, Mohaupt M, Klimkait T. Prospective monitoring of BK virus load after discontinuing sirolimus treatment in a renal transplant patient with BK virus nephropathy. J Infect Dis. 2001 Dec 1;184(11):1494-5; author reply 1495-6. doi: 10.1086/324425. No abstract available. PMID 11709797
- [Background] Binet I, Nickeleit V, Hirsch HH, Prince O, Dalquen P, Gudat F, Mihatsch MJ, Thiel G. Polyomavirus disease under new immunosuppressive drugs: a cause of renal graft dysfunction and graft loss. Transplantation. 1999 Mar 27;67(6):918-22. doi: 10.1097/00007890-199903270-00022. PMID 10199744
- [Background] Weimer R, Susal C, Yildiz S, Streller S, Pelzl S, Staak A, Renner F, Dietrich H, Daniel V, Feuring E, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. sCD30 and neopterin as risk factors of chronic renal transplant rejection: impact of cyclosporine A, tacrolimus, and mycophenolate mofetil. Transplant Proc. 2005 May;37(4):1776-8. doi: 10.1016/j.transproceed.2005.02.088. PMID 15919463
- [Background] Weimer R, Staak A, Susal C, Streller S, Yildiz S, Pelzl S, Renner F, Dietrich H, Daniel V, Rainer L, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. ATG induction therapy: long-term effects on Th1 but not on Th2 responses. Transpl Int. 2005 Feb;18(2):226-36. doi: 10.1111/j.1432-2277.2004.00047.x. PMID 15691277
- [Background] Weimer R, Mytilineos J, Feustel A, Preiss A, Daniel V, Grimm H, Wiesel M, Opelz G. Mycophenolate mofetil-based immunosuppression and cytokine genotypes: effects on monokine secretion and antigen presentation in long-term renal transplant recipients. Transplantation. 2003 Jun 27;75(12):2090-9. doi: 10.1097/01.TP.0000058808.37349.23. PMID 12829918
- [Background] Weimer R, Streller S, Staak A, Heilke M, Li D, Dietrich H, Daniel V, Feustel A, Rainer L, Zinn S, Friemann S, Ernst W, Grimm H, Padberg W, Zimmermann T, Opelz G. Effects of three immunosuppressive regimens on CD4 helper function, B cell monocyte and cytokine responses in renal transplant recipients: 4-month follow-up of a prospective randomized study. Transplant Proc. 2002 Sep;34(6):2377-8. doi: 10.1016/s0041-1345(02)03278-5. No abstract available. PMID 12270445
- [Background] Weimer R, Melk A, Daniel V, Friemann S, Padberg W, Opelz G. Switch from cyclosporine A to tacrolimus in renal transplant recipients: impact on Th1, Th2, and monokine responses. Hum Immunol. 2000 Sep;61(9):884-97. doi: 10.1016/s0198-8859(00)00152-x. PMID 11053632
- [Background] Daniel V, Arzberger J, Melk A, Weimer R, Ruhenstroth A, Carl S, Wiesel M, Opelz G. Predictive indicators of rejection or infection in renal transplant patients. Transplant Proc. 1999 Feb-Mar;31(1-2):1364-5. doi: 10.1016/s0041-1345(98)02030-2. No abstract available. PMID 10083605
- [Background] Weimer R, Zipperle S, Daniel V, Carl S, Staehler G, Opelz G. Pretransplant CD4 helper function and interleukin 10 response predict risk of acute kidney graft rejection. Transplantation. 1996 Dec 15;62(11):1606-14. doi: 10.1097/00007890-199612150-00014. PMID 8970616
- [Background] Daniel V, Pasker S, Wiesel M, Carl S, Pomer S, Staehler G, Schnobel R, Weimer R, Opelz G. Cytokine monitoring of infection and rejection in renal transplant recipients. Transplant Proc. 1995 Feb;27(1):884-6. No abstract available. PMID 7879219
- [Background] Weimer R, Zipperle S, Daniel V, Pomer S, Staehler G, Opelz G. IL-6 independent monocyte/B cell defect in renal transplant recipients with long-term stable graft function. Transplantation. 1994 Jan;57(1):54-9. doi: 10.1097/00007890-199401000-00011. PMID 7507271
- [Background] Weimer R, Daniel V, Zimmermann R, Schimpf K, Opelz G. Autoantibodies against CD4 cells are associated with CD4 helper defects in human immunodeficiency virus-infected patients. Blood. 1991 Jan 1;77(1):133-40. PMID 1824617
- [Background] Weimer R, Daniel V, Pomer S, Opelz G. B lymphocyte response as an indicator of acute renal transplant rejection. II. Pretransplant and posttransplant B cell responses of m mitogen and donor cell-stimulated cultures. Transplantation. 1989 Oct;48(4):572-5. PMID 2678634
- [Background] Weimer R, Daniel V, Pomer S, Opelz G. B lymphocyte response as an indicator of acute renal transplant rejection. I. Immunoglobulin-secreting cells in peripheral blood. Transplantation. 1989 Oct;48(4):569-72. PMID 2572082
- [Background] Susal C, Dohler B, Opelz G. Graft-protective role of high pretransplantation IgA-anti-Fab autoantibodies: confirmatory evidence obtained in more than 4000 kidney transplants. The Collaborative Transplant Study. Transplantation. 2000 Apr 15;69(7):1337-40. doi: 10.1097/00007890-200004150-00021. PMID 10798750
- [Background] Pelzl S, Opelz G, Daniel V, Wiesel M, Susal C. Evaluation of posttransplantation soluble CD30 for diagnosis of acute renal allograft rejection. Transplantation. 2003 Feb 15;75(3):421-3. doi: 10.1097/01.TP.0000044702.18327.66. PMID 12589170
- [Background] Susal C, Pelzl S, Dohler B, Opelz G. Identification of highly responsive kidney transplant recipients using pretransplant soluble CD30. J Am Soc Nephrol. 2002 Jun;13(6):1650-6. doi: 10.1097/01.asn.0000014256.75920.5b. PMID 12039995
- [Background] Susal C, Opelz G. Kidney graft failure and presensitization against HLA class I and class II antigens. Transplantation. 2002 Apr 27;73(8):1269-73. doi: 10.1097/00007890-200204270-00014. PMID 11981420